CLINICAL TRIAL: NCT02063984
Title: Behavioral Treatment of Adolescent Marijuana Use
Brief Title: Behavioral Treatment of Adolescent Substance Use
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Mountain Manor Treatment Center (Other); University of Pennsylvania (Other); Johns Hopkins University (Other); Spectrum Youth and Family Services (Other)
Responsible Party: Principal Investigator, Alan J. Budney, Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA015186-DartmouthSpectrum; R01DA015186-12A1 (NIH)
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Results first posted 2021-05-10 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Outpatient Treatment (IOP) + Contingency Management (CM) + Working Memory Training (WMT) (Experimental): IOP + CM + WMT
  Interventions: Behavioral: Intensive Outpatient Treatment (IOP) + Contingency Management (CM); Behavioral: Working Memory Training
- IOP + CM (Active Comparator): IOP + CM
  Interventions: Behavioral: Intensive Outpatient Treatment (IOP) + Contingency Management (CM)

INTERVENTIONS:
Behavioral: Intensive Outpatient Treatment (IOP) + Contingency Management (CM) — Multiple group sessions weekly, one individual counseling session weekly with teen to review and discuss contingency management abstinence-based incentives
Behavioral: Working Memory Training — 25 computer-delivered sessions of neurocognitive training
  Other Names: Cogmed, Inc
  Arms: Intensive Outpatient Treatment (IOP) + Contingency Management (CM) + Working Memory Training (WMT)

SUMMARY:
This study will continue research designed to improve treatment outcomes for adolescent substance use disorders by integrating neuroscience- and behaviorally-based treatments. In particular, this project will be the first to evaluate whether Working Memory Training can enhance cognitive function and reduce impulsive decision making to improve abstinence outcomes. In addition, an adaptive abstinence-based incentive program will be evaluated as a new method for intervening with those who do not respond to their first-line treatment.

DETAILED DESCRIPTION:
The study will test two novel strategies to enhance outcomes. Working Memory Training (WMT), an efficacious method for strengthening specific cognitive processes, aims to improve factors (e.g., delay discounting / impulsive decision-making) that have shown a strong relation to substance use and treatment response. Second, more intensive and higher magnitude CM (ICM) will be used to motivate abstinence among teens who are not abstinent by Week 4. The investigators hypothesize that these strategies will improve outcomes by modifying a fundamental cognitive system involved in making choices to engage in risky behavior and by increasing motivation to abstain in early nonresponders. Aim 1 will pilot and refine the new procedures in a community clinic in preparation for the randomized trial. A sequential, multiple assignment randomized trial (SMART) will allow the study to determine the most effective first-line treatment and the most effective adaptive strategy (Aim 2). All teens will begin treatment with CM or CM/WMT. After 4 weeks, responders will continue in their first-line treatments, while nonresponders will be randomized to ICM or to continue with first-line treatment. Aim 3 will conduct mechanistic analyses to assess whether cognitive changes related to WMT engender increased abstinence, and whether specific tailoring variables moderate treatment effects. Aim 4 will gather formative data on implementation factors to inform future large-scale studies and dissemination efforts. Primary hypotheses are: (1) first-line treatment with WMT will improve abstinence outcomes and reduce relapse; (2) strategies with ICM for nonresponders will result in better outcomes than those without; (3) WMT will reduce delay discounting, which will predict outcome. The unique approach holds promise for reducing multiple types of risky behaviors by affecting basic mechanisms that determine impulsive decision-making.

ELIGIBILITY:
Inclusion Criteria:

Participants must be 12 to 26 years of age, must live at home with the parent who will participate, report using marijuana during the previous 30 days or provide a marijuana-positive urine test, meet criteria for cannabis abuse or dependence, and have a parent who can participate.

Exclusion Criteria: DSM criteria for dependence (likely to be adjusted for DSM-5 Use Disorder) on alcohol or other drugs other than marijuana (use of or meeting criteria for abuse of other substances will not be an exclusion criterion), active psychosis, severe medical or psychiatric illness limiting participation, or pregnant or breast-feeding.

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Budney, Ph.D, Principal Investigator — Dartmouth College
Locations (1):
- Mountain Manor Treatment Center, Baltimore, Maryland, United States

REFERENCES:
- [Result] Stanger C, Scherer EA, Vo HT, Babbin SF, Knapp AA, McKay JR, Budney AJ. Working memory training and high magnitude incentives for youth cannabis use: A SMART pilot trial. Psychol Addict Behav. 2020 Feb;34(1):31-39. doi: 10.1037/adb0000480. Epub 2019 Jun 27. PMID 31246068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from a community intensive outpatient program from December 2015 to October 2017.
Groups:
- CM + WMT: Intensive Outpatient Treatment + Contingency Management + Working Memory Training (IOP + CM + WMT)
- CM + No WMT: Intensive Outpatient Treatment + Contingency Management (IOP + CM)
Period: Overall Study
Arm/Group | CM + WMT | CM + No WMT
Started | 29 | 30
Completed | 23 | 25
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CM + WMT | CM + No WMT | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.0 (1.5) | 16.7 (2.1) | 16.35 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 21 | 21 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 26 | 28 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 24 | 45
  White | 8 | 4 | 12
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Any Cannabis Abstinence
Description: Number of participants with any cannabis abstinence during treatment
Time Frame: Intervention weeks 1 to 14
Population: Participants who met Cannabis Use Disorder criteria, excluding those who met other drug use disorder criteria.
Measure: Number; unit: participants
Arm/Group | CM + WMT | CM + No WMT
Number analyzed (Participants) | 29 | 30
participants | 13 | 18
Statistical Analysis 1: Comparison: CM + WMT vs CM + No WMT; CM+No WMT is the comparison condition; Test type: Superiority; Odds Ratio (OR) = .42, 95% CI 2-sided [.11 to 1.56] — Outcome was tested in a zero-inflated negative binomial (ZINB) model

2. Primary Outcome: Weeks of Continuous Cannabis Abstinence
Description: Weeks of continuous abstinence during treatment
Time Frame: 14 week treatment period
Population: Calculated only for those who achieved at least one week of abstinence during the treatment period
Measure: Mean (Standard Deviation); unit: Weeks of Continuous Abstinence
Arm/Group | CM + WMT | CM + No WMT
Number analyzed (Participants) | 13 | 18
Weeks of Continuous Abstinence | 7.15 (4.63) | 4.88 (4.35)
Statistical Analysis 1: Comparison: CM + WMT vs CM + No WMT; CM+No WMT is the comparison condition; Test type: Superiority; Ratio of means = 1.56, 95% CI 2-sided [.79 to 3.07] — Outcome was tested in a zero-inflated negative binomial (ZINB) model

3. Secondary Outcome: Any Days of Cannabis Use
Description: Number of participants with any days of cannabis use during treatment
Time Frame: Intervention weeks 1 to 14
Population: Participants with Cannabis Use Disorder and with non-missing data on 25% or more of treatment days (excluding those with other drug use disorder)
Measure: Count of Participants; unit: Participants
Arm/Group | CM + WMT | CM + No WMT
Number analyzed (Participants) | 18 | 19
Participants | 11 | 14
Statistical Analysis 1: Comparison: CM + WMT vs CM + No WMT; CM+No WMT is the comparison condition; Test type: Superiority; Odds Ratio (OR) = .93, 95% CI 2-sided [.18 to 4.82]

4. Secondary Outcome: Days of Cannabis Use
Description: Percent of Days Used During the Treatment Period
Time Frame: The intervention period between Week 1 and Week 14
Measure: Mean (Standard Deviation); unit: percentage of days of cannabis use
Arm/Group | CM + WMT | CM + No WMT
Number analyzed (Participants) | 11 | 14
percentage of days of cannabis use | 32.5 (31.0) | 24.5 (23.3)
Statistical Analysis 1: Comparison: CM + WMT vs CM + No WMT; CM+No WMT is the comparison condition; Test type: Superiority; Ratio of means = .92, 95% CI 2-sided [.33 to 2.54] — Outcome was tested in a zero-inflated negative binomial (ZINB) model

5. Secondary Outcome: Any Cannabis Abstinence Across Four Treatment Strategies
Description: Number of participants who achieved at least one week of abstinence
Time Frame: Treatment period between week 1 and week 14
Population: Ns in each strategy are the sum of [1] dropouts in the phase 1 condition, [2] responders in the phase 1 condition; and [3] nonresponders in the phase 1 condition who are assigned to the specified phase 2 condition. These ns for each strategy are: [1] 5+8+8=21; [2] 6+10+5=21; [3] 5+8+8=21; [4] 6+10+8=24.
Measure: Count of Participants; unit: Participants
Groups:
- Strategy 1: Start in CM stay in CM
- Strategy 2: Start in CM+WMT stay in CM+WMT
- Strategy 3: Start in CM responders stay in CM, non-responders get Enhanced CM
- Strategy 4: Start in CM+WMT responders stay in CM+WMT, non-responders get Enhanced CM+WMT
Arm/Group | Strategy 1 | Strategy 2 | Strategy 3 | Strategy 4
Number analyzed (Participants) | 21 | 21 | 21 | 24
Participants | 12 | 12 | 14 | 11
Statistical Analysis 1: Comparison: Strategy 1 vs Strategy 2; Strategy 1 is the comparison condition; Test type: Superiority; Odds Ratio (OR) = 1.04, 95% CI 2-sided [.45 to 2.45]
Statistical Analysis 2: Comparison: Strategy 1 vs Strategy 3; Strategy 1 is the comparison condition; Test type: Superiority; Odds Ratio (OR) = 2.29, 95% CI 2-sided [.84 to 6.20]
Statistical Analysis 3: Comparison: Strategy 1 vs Strategy 4; Strategy 1 is the comparison condition; Test type: Superiority; Odds Ratio (OR) = .51, 95% CI 2-sided [.23 to 1.13]

6. Secondary Outcome: Weeks of Cannabis Abstinence Across Four Treatment Strategies
Description: Mean weeks of continuous cannabis abstinence among those who achieved at least one week of abstinence
Time Frame: Treatment period between week 1 and week 14
Population: Participants with at least one week of cannabis abstinence during treatment
Measure: Mean (Standard Deviation); unit: weeks of continuous abstinence
Arm/Group | Strategy 1 | Strategy 2 | Strategy 3 | Strategy 4
Number analyzed (Participants) | 12 | 12 | 14 | 11
weeks of continuous abstinence | 6.17 (4.73) | 7.42 (4.74) | 5.29 (4.43) | 7.82 (4.75)
Statistical Analysis 1: Comparison: Strategy 1 vs Strategy 2; Strategy 1 is the comparison condition; Test type: Superiority; Ratio of means = 1.21, 95% CI 2-sided [.76 to 1.92]
Statistical Analysis 2: Comparison: Strategy 1 vs Strategy 3; Strategy 1 is the comparison condition; Test type: Superiority; Ratio of means = .76, 95% CI 2-sided [.49 to 1.18]
Statistical Analysis 3: Comparison: Strategy 1 vs Strategy 4; Strategy 1 is the comparison condition; Test type: Superiority; Ratio of means = 1.33, 95% CI 2-sided [.83 to 2.15]

ADVERSE EVENTS:
Time Frame: Information will be collected from the scheduled first study visit through the 12 month follow-up assessment visit. (12 months total)
Arm/Group | Intensive Outpatient Treatment (IOP) + Contingency Management (CM) + Working Memory Training (WMT) | IOP + CM
All-Cause Mortality (participants affected / at risk) | 2/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 8/29 | 7/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Outpatient Treatment (IOP) + Contingency Management (CM) + Working Memory Training (WMT) (N=29) | IOP + CM (N=30)
Overdose (Psychiatric disorders) | 2 (2) | 0 (0)
Suicidal ideation without a plan (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Incarceration (Social circumstances) | 3 (3) | 4 (4)
Arrest (Social circumstances) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Drug induced psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT02063984/Prot_SAP_000.pdf